CLINICAL TRIAL: NCT03580291
Title: A Randomized, Double-Blind, Parallel-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Human Umbilical Cord Mesenchymal Stem Cells in Patients With Lupus Nephritis
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells Treatment for Lupus Nephritis (LN)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lingyun Sun (Other)
Responsible Party: Sponsor-Investigator, Lingyun Sun, Director of Department of Rheumatology and Immunology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017001
Record Dates: First submitted 2018-01-12; First posted 2018-07-09 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; Mesenchymal stem cell
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): The group receive pulse infusion of MSCs and placebo of oral Mycophenolate Mofetil (MMF). The cells of 2 x 10^6/kg body weight are suspended in 100ml saline and infused intravenously.
  1. Dexamethasone of 10mg is intravenously injected before 30 minutes of cells infusion.
  2. A sterile blood transfusion device is used during the venous transfusion, and it is washed with saline before infusion. Take a slow infusion of about 20 drops per minute in the first 15 minutes. Increase to about 60 drops per minute if the patient had no complaints of discomfort.
  Interventions: Other: Mesenchymal stem cells; Drug: Placebo of Mycophenolate Mofetil
- Mycophenolate Mofetil (Active Comparator): The group receive placebo of MSCs and oral Mycophenolate Mofetil of 2.0g/d. .
  Interventions: Drug: Mycophenolate Mofetil; Other: Placebo of Mesenchymal stem cells

INTERVENTIONS:
Other: Mesenchymal stem cells — The group receive pulse infusion of MSCs once of 2 x 10^6/kg body weight
  Arms: Mesenchymal stem cells
Drug: Mycophenolate Mofetil — This group receive oral MMF of 2.0 g / d.
  Arms: Mycophenolate Mofetil
Other: Placebo of Mesenchymal stem cells — The group receive placebo of Mesenchymal stem cells.
  Arms: Mycophenolate Mofetil
Drug: Placebo of Mycophenolate Mofetil — The group receive placebo of oral mycophenolate mofetil.
  Arms: Mesenchymal stem cells

SUMMARY:
Lupus nephritis (LN) is one of the most serious complications and the main cause of death in patients with systemic lupus erythematosus (SLE).The investigators have investigated the usefulness, and confirmed the efficacy and safety of mesenchymal stem cells (MSC) treatment of LN in animal models, in vitro experiments and phase I clinical trial. In this study, a randomized, placebo-controlled, parallel group, non-inferiority, prospective, multicenter clinical trial is performed to investigate the efficacy and safety of MSC transplantation in the treatment of LN compared to mycophenolate mofetil (MMF).

DETAILED DESCRIPTION:
Lupus nephritis (LN) is one of the most serious complications and the main cause of death in patients with systemic lupus erythematosus (SLE). Type III, type IV and type V LN are severe clinical entities with poor prognosis, and its treatment remains challenging. Currently, type III, type IV, type V, type III plus V and type IV plus V LN are treated mainly according to the guidelines developed by KDIGO and the European Association for Anti-Rheumatism and European League Against Rheumatism/European Renal Association-European Dialysis and Transplant Association (EULAR/ERAEDTA). The main therapeutic regimens recommended by these guidelines include glucocorticoid combined with immunosuppressants such as cyclophosphamide (CTX), mycophenolate mofetil (MMF), etc. These medications can significantly induce disease remission and improve the long-term survival. However, some patients do not adequately response to the treatment of the combination of steroids and immunosuppressants, and the disease activity cannot be well-controlled. The high prevalence of steroids and immunosuppressants related adverse effects, such as steroid-related diabetes, bone necrosis, hypertension, peptic ulcer, CTX-related bone marrow and gonadal suppression, MMF-related infection risk and so on, have been found in long-term follow-up study. In addition, to date, there is insufficient data to support the use of new biologics, such as rituximab and abatacept in the induction therapy in patients with LN.

Mesenchymal stem cells (MSCs) can be obtained from several tissues and possess multiple differentiation potencies and immunomodulatory effects. The investigators have investigated the usefulness, and confirmed the efficacy and safety of MSC treatment of LN in animal models, in vitro experiments and phase I clinical trial. The studies also for the first time found that the MSC abnormalities are involved in the onset and development of lupus both in the lupus mice model and in SLE patients. The investigators found that the efficacy of allogeneic (xenogeneic) MSC transplantation is superior to autologous MSC transplantation in LN mice model. Thus, in current opinion, SLE is not only a hematopoietic stem cell disease, but also a mesenchymal stem cell disease. The investigators treated the refractory LN patients with allogenic MSC treatment, the outcomes revealed that the total response rate was 60%, the mortality rate of 2 to 5 years decreased from 35% - 45% to 6%. These results strongly support the use of allogenic MSC transplantation in the refractory LN patients. The mechanisms of MSC treatment include correcting the immune unbalance, inducing immune tolerance, tissue repair and the improvement of organ function. Allogeneic MSC transplantation for the treatment of SLE and other refractory autoimmune diseases have shown significant efficacy and excellent safety. However, these studies have limitations due to the lack of large-scale, multi-center, randomized, controlled, prospective study to further confirm the efficacy of allogeneic MSC transplantation, as well as the guideline for MSC treatment in SLE needs to be developed. Therefore, a randomized, placebo-controlled, parallel group, non-inferiority, prospective, multicenter clinical trial is urgent needed to promote the application of MSC transplantation in SLE treatment, to bring the benefit of the patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who met the American college of Rheumatology (ACR, 1997) classification criteria for SLE;
2. Ages: 18-60 years old (including);
3. Presence of class III, IV, V, III+V or IV+V LN as determined by renal biopsy within 12 weeks of randomization(2003 ISN/RPS LN classification criteria);
4. Morning proteinuria /creatinine ratio >1.0 or 24 hours Proteinuria >1.0g, with or without microscopic hematuria(>5 red blood cells/high-power field);
5. Women of childbearing age agreed to adopt effective contraception measures during the trial period;
6. Urine pregnancy tests were negative in women of childbearing age;
7. Subject signed the informed consent form voluntarily and complied with the requirements of the research program.

Exclusion Criteria:

1. Received MMF, CTX, other potent immunosuppressive agents (including cyclosporine, tacrolimus, Tripterygium wilfordii and leflunomide) or biologics (Rituximab or others) within the past 12 weeks.
2. Previous failure to respond to MMF.
3. Known intolerance to MMF.
4. Renal biopsy showing ≥50% glomerulus sclerosis.
5. Renal biopsy showing capillary loops necrosis, microthrombus formation in capillary loops, or cellular crescent in ≥50% of glomeruli.
6. Patients diagnosed with other autoimmune diseases apart from SLE: dermatomyositis/polymyositis, mixed connective tissue disease, scleroderma, rheumatoid arthritis, etc. However, participants with secondary Sjogren's syndrome are allowed to take part in the study.
7. Patients suffering from severe liver or kidney dysfunction (total bilirubin more than 14mg/L, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal lab value; creatinine clearance rate (Ccr) < 30ml/min or serum creatinine (Scr) ≥265.2umol/L).
8. Patients with hematological abnormalities (white blood cell <3000/uL, hemoglobin <8g/dL, and/or platelets <50000/uL).
9. Patients diagnosed with severe or uncontrolled cardiovascular, neurological, pulmonary (including obstructive pulmonary disease and interstitial lung disease), hepatic, endocrine (including uncontrolled diabetes mellitus), and gastrointestinal disorders.
10. Known active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis, atypical mycobacterial infection, granulomatous disease showed by chest X-ray, hepatitis B, hepatitis C, HIV infection and herpes zoster, whereas not including onychomycosis). Any infection requiring hospitalization within 4 weeks prior to enrollment or intravenous antimicrobial treatment within 2 weeks prior to randomization.
11. History of malignancy, including solid tumor and hematologic malignancies (except basal cell carcinoma which has been excised or successfully treated).
12. Women who are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Total remission rate | weeks 24
  Complete remission rate (CR) and partial remission rate (PR)

SECONDARY OUTCOMES:
The time for subjects of the two groups to achieve PR and CR | Baseline to weeks 24
Levels of 24-hour urinary protein | Baseline, weeks 4, 8, 12, 16, 20, 24
Ratio of Urinary Protein / Creatinine | Baseline, weeks 4, 8, 12, 16, 20, 24
Levels of serum albumin | Baseline, weeks 4, 8, 12, 16, 20, 24
Levels of serum creatinine | Baseline, weeks 4, 8, 12, 16, 20, 24
The estimated glomerular filtration rate ( eGFR ) | Baseline, weeks 4, 8, 12, 16, 20, 24
Levels of Complement component 3 (C3) | Baseline, weeks 4, 8, 12, 16, 20, 24
Levels of Complement component 4 (C4) | Baseline, weeks 4, 8, 12, 16, 20, 24
The antinuclear antibody (ANA) levels | Baseline, weeks 4, 8, 12, 16, 20, 24
The anti-double stranded DNA antibody (dsDNA) levels | Baseline, weeks 4, 8, 12, 16, 20, 24
Patient Health Assessment Questionnaire (HAQ) score | Baseline, weeks 4, 8, 12, 16, 20, 24
Physician Global Assessment (PhGA) score | Baseline, weeks 4, 8, 12, 16, 20, 24
The (Systemic lupus Erythematosis Disease Activity index) SLEDAI score | Baseline, weeks 4, 8, 12, 16, 20, 24
The (British Isles lupus assessment group ) BILAG score | Baseline, weeks 4, 8, 12, 16, 20, 24
The SLE reaction index | Baseline, weeks 4, 8, 12, 16, 20, 24
Total remission rate | weeks 12
  Complete remission rate (CR) and partial remission rate (PR)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to weeks 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided